CLINICAL TRIAL: NCT05426070
Title: Preliminary Efficacy of a Strength Training Intervention on Exercise Adherence and Weight Among Pre-Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 580913
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Physical Inactivity; Obesity
Keywords: strength training; group-based exercise; pre-menopausal; exercise adherence
MeSH Terms: conditions — Sedentary Behavior; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength training-based exercise (Experimental): The strength training-based exercise intervention will be delivered via group-based Zoom sessions, motivational text messages, and a website. Participants will take part in two group-based Zoom exercise sessions (40-minute exercise sessions and 20 minutes of motivational counseling) and two individual exercise sessions per week for three months. Exercise sessions will include a combination of various aerobic and muscle strengthening exercises designed to keep heart rate in the 60-85% range of maximum heart rate. Motivational counseling will be focused on increasing motivation to exercise and habit formation. Strength training-based participants will also receive access to a mobile phone-friendly study website and will receive email messages. Both the website and email messages will contain motivational content to complete the exercise sessions.
  Interventions: Behavioral: Strength training-based exercise
- No contact, wait-list control (No Intervention): Participants in the no contact, wait-list control intervention will participate in assessments at baseline and three months. Following the six month assessment, participants will have the option of receiving the strength training-based intervention as described above.

INTERVENTIONS:
Behavioral: Strength training-based exercise — Participants will take part in two group-based Zoom exercise sessions and two individual exercise sessions per week for three months. Exercise sessions will include a combination of various aerobic (e.g., jogging in place, high knees) and muscle strengthening exercises (e.g., burpees, push-ups, lunges, body weight squats) designed to keep heart rate in the 60-85% range of maximum heart rate. Participants will choose from a variety of options for their two individual sessions (e.g., online exercise video, jogging or walking outside, prescribed exercise session listed on the website, or any other exercise) and modifications for each exercise will be made depending on the participant's ability and current fitness and strength level. Participants will be instructed to stop exercising if problems occur and will receive training and handouts on how to recognize problems such as angina and myocardial infarction.
  Arms: Strength training-based exercise

SUMMARY:
The purpose of this study is to examine the feasibility and acceptability of a strength training-based intervention on exercise adherence among low active (defined as engaging in physical activity 90 minutes or less per week), pre-menopausal women ages 40-50, along with the effect on weight and various psychosocial measures. Participants will be randomly assigned to a strength training-based intervention or a wait-list control each lasting three months (participants in the no contact, wait-list control condition will have the option of receiving the strength training-based intervention following the three months).

DETAILED DESCRIPTION:
Participants will be randomly assigned to a strength training-based exercise intervention or a no contact, wait-list control each lasting three months (participants in the no contact, wait-list control will have the option of receiving the strength training-based intervention following the three months). The strength training-based exercise intervention will be delivered via group-based Zoom sessions, motivational email messages, and a website. Participants will take part in two group-based Zoom exercise sessions (40-minute exercise sessions and 20 minutes of motivational counseling) and two individual exercise sessions per week for six months. Exercise sessions will include a combination of various aerobic (e.g., jogging in place, high knees) and muscle strengthening exercises (e.g., burpees, push-ups, lunges, body weight squats) designed to keep heart rate in the 60-85% range of maximum heart rate. Participants will choose from a variety of options for their two individual sessions (e.g., online exercise video, jogging or walking outside, prescribed exercise session listed on the website, or any other exercise) and modifications for each exercise will be made depending on the participant's ability and current fitness and strength level (e.g., wall push-ups vs. knee push-ups vs. regular push-ups). Participants will be instructed to stop exercising if problems occur and will receive training and handouts on how to recognize problems such as angina and myocardial infarction symptoms.

Self-Determination Theory (SDT) and habit formation theory will guide the content of the counseling portion of the Zoom sessions and the motivational features of the study website and text messages. Motivational counseling will be focused on increasing motivation to exercise and habit formation. The goal is to achieve integrated regulation and therefore, the health counselor will focus on positive affective response to exercise sessions and discuss how being physically active is becoming part of their self-identity. The goal will be high intrinsic motivation (i.e., individuals engage in exercise due to inherent pleasure) since it is related to higher levels of exercise. Strength training-based participants will also receive access to a mobile phone-friendly study website and will receive emails. Both the website and email messages will contain motivational content to complete the exercise sessions. The motivational website will also include an online log to track completion of home-based sessions and options for individual-based exercise sessions.. Assessment of exercise adherence, weight, and psychosocial variables will occur at baseline and three months.

ELIGIBILITY:
Inclusion Criteria:

* 1) pre-menopausal women ages 40-50 years; (2) engaging in 90 minutes or less of exercise per week; (3) no exercise contraindications; (4) adequate space at home to complete exercise sessions and capacity to use Zoom via a mobile device or computer; (5) available to attend two zoom-based sessions a week; (6) be able to read, understand, and speak in the English language (7) willing to be randomly assigned to either study condition (8) access to iPhone 8 or later with iOS 16 or later

Exclusion Criteria:

* Specific exclusion criteria will include a history of coronary heart disease (history of myocardial infarction, symptoms of angina), orthopedic problems that would limit physical activity participation, diabetes, stroke, osteoarthritis, and any other medical condition that may make physical activity unsafe or unwise. Other exclusion criteria will include current or planned pregnancy, psychosis or current suicidal ideation, and psychiatric hospitalization within the last six months.

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 39 (Actual)
Dates: Start 2022-12-30 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Exercise Adherence | from date of randomization until the date of three month assessment; up to three months
  Apple Watch

SECONDARY OUTCOMES:
Weight | from date of randomization until the date of three month assessment; up to three months
  Withings Smart Scale

OTHER OUTCOMES:
Physical Activity Enjoyment Scale (PACES) | from date of randomization until the date of three month assessment; up to three months
  questionnaire; Physical Activity Enjoyment Scale (PACES) is an 18 item scale that assesses enjoyment for physical activity by asking participants to rate "how you feel at the moment about the physical activity you have been doing" using a 7-point bipolar Likert scale from 1 (I enjoy it) to 7 (I hate it). Higher scores indicate higher enjoyment with range of 18-126 being possible.
Behavioral Regulation in Exercise Questionnaire (BREQ-2) | from date of randomization until the date of three month assessment; up to three months
  questionnaire; the Behavioral Regulation in Exercise Questionnaire (BREQ-2) is a 19-item questionnaire that includes five subscales (intrinsic motivation, identified regulation, introjected regulation, external regulation, and amotivation. This scale is on a 5 point Likert scale ranging from 0 (not true for me) to 4 (very true for me). The minimum score is -24 and the maximum score is +20. Higher positive scores indicate more autonomous motivation whereas lower negative scores indicate less autonomous motivation.
Motives for Physical Activity Measure- Revised (MPAM-R) | from date of randomization until the date of three month assessment; up to three months
  questionnaire; the Motives for Physical Activity Measure- Revised (MPAM-R) is a 30-item scale that examines five motives for physical activity participation including enjoyment/interest, competence/challenge, social interaction, appearance, and fitness. Composed of 30 items, 7-point Likert scale with 1= not at all true for me to 7= very true for me. Maximum score=210; minimum score=30. Higher score=higher motivation.
Physical Activity Self-Efficacy | from date of randomization until the date of three month assessment; up to three months
  questionnaire; physical activity self-efficacy measuring how confident of exercise. 5 items. 5-point Likert scale with 1=not at all confident to 5= extremely confident. Maximum value of 25, minimum value of 5 with higher scores indicating higher level of self-efficacy
Outcome Expectations or Exercise | from date of randomization until the date of three month assessment; up to three months
  questionnaire; Outcome Expectations for Exercise measures the degree to which individuals agree to statements regarding benefits of exercise. 9 items. 5-point Likert scale with 1= strongly disagree to 5= strongly agree. Maximum value= 45; minimum value= 9 with higher score indicating higher outcome expectations related to exercise.
Social Support for Physical Activity | from date of randomization until the date of three month assessment; up to three months
  questionnaire; Social Support for Physical Activity measures perceived social support based on two subscales; family and friends. 13 items. 5-point Likert scale with 0=none and 4=very often. Maximum score= 52; minimum score=0. Higher levels indicate higher level of perceived social support for physical activity.
Exercise Feeling Inventory Survey | from date of randomization until the date of three month assessment; up to three months
  questionnaire; Exercise Feeling Inventory Survey (EFI) measures feeling states that occur during acute PA bouts. Four feeling states are assessed including revitalization, positive engagement, physical exhaustion, and tranquility. 12 items. 5-point Likert scale; 0= do not feel and 4=feel very strongly. Maximum Score= 48; minimum score=0. Higher score= higher feeling.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ryan, R. M., & Deci, E. L. (2002). Overview of self-determination theory: An organismic dialectical perspective. Handbook of Self-determination Research, 2, 3-33.
- [Background] Lally P, Wardle J, Gardner B. Experiences of habit formation: a qualitative study. Psychol Health Med. 2011 Aug;16(4):484-9. doi: 10.1080/13548506.2011.555774. PMID 21749245
- [Background] Thogersen-Ntoumani C, Shepherd SO, Ntoumanis N, Wagenmakers AJ, Shaw CS. Intrinsic motivation in two exercise interventions: Associations with fitness and body composition. Health Psychol. 2016 Feb;35(2):195-8. doi: 10.1037/hea0000260. Epub 2015 Sep 21. PMID 26389719
- [Derived] Lewis BA, Schuver KJ, Swinney KB, Dregney TM, Linde JA. Examining the feasibility and preliminary efficacy of a group-based physical activity intervention integrating strength training among pre- and perimenopausal women: A randomized pilot trial. Womens Health (Lond). 2025 Jan-Dec;21:17455057251361243. doi: 10.1177/17455057251361243. Epub 2025 Aug 10. PMID 40784014